CLINICAL TRIAL: NCT05610631
Title: Swiss PH Registry - Cohort of Swiss PH Patients
Brief Title: Pulmonary Hypertension Registry Switzerland
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Actelion (Industry)
Responsible Party: Sponsor
Other Study IDs: Swiss PH Registry
Record Dates: First submitted 2022-11-01; First posted 2022-11-09 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Pulmonary arterial hypertension: Pulmonary arterial hypertension
- PH due to left heart diseases: PH due to left heart diseases
- PH due to lung disease and/or hypoxia: PH due to lung disease and/or hypoxia
- Chronic thromboembolic PH: Chronic thromboembolic PH
- Miscellaneous PH: Miscellaneous PH

SUMMARY:
Registry Data from PH-patients in Switzerland, who have given consent to records for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PH

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pulmonary Hypertension (PH)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
6-minute walking distance | within the study duration e.g. up to 10 years
  6-minute walking distance

SECONDARY OUTCOMES:
New York Heart Association functional class | within the study duration e.g. up to 10 years
  New York Heart Association functional class
NTproBNP | within the study duration e.g. up to 10 years
  NTproBNP
Survival | within the study duration e.g. up to 10 years
  time to death analysis
Medication | within the study duration e.g. up to 10 years
  escalation of clinical therapy

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich, Prof. Dr., Principal Investigator — UniversityHospital Zurich
Locations (1):
- Respiratory Clinic, University Hospital of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No